CLINICAL TRIAL: NCT02212561
Title: A Phase I/II Study of the Selective Inhibitor of Nuclear Export Selinexor (KPT-330) in Combination With Fludarabine and Cytarabine in Patients With Refractory or Relapsed Leukemia or Myelodysplastic Syndrome
Brief Title: Selinexor With Fludarabine and Cytarabine for Treatment of Refractory or Relapsed Leukemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SELHEM; NCI-2014-01704 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2014-07-30; First posted 2014-08-08 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2017-02

CONDITIONS: Acute Myeloid Leukemia (AML); Acute Lymphoblastic Leukemia (ALL); Myelodysplastic Syndrome (MDS); Mixed Phenotype Acute Leukemia (MPAL)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Leukemia, Biphenotypic, Acute | interventions — selinexor; fludarabine; fludarabine phosphate; Cytarabine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Interventions: Selinexor, Fludarabine, and Cytarabine. Methotrexate/hydrocortisone/cytarabine (intrathecal triples) will be given prior to cycle 1.
  Interventions: Drug: Selinexor; Drug: Fludarabine; Drug: Cytarabine; Drug: methotrexate/hydrocortisone/cytarabine

INTERVENTIONS:
Drug: Selinexor — Given orally on days 1,3,8,10,22 and 24 of each cycle
  Other Names: KPT-330
Drug: Fludarabine — Will be given intravenously (IV) over 30 minutes daily on days 16 through 20. Fludarabine may be given prior to day 16 if it is determined to be in the participant's best interest based on disease progression. Chemotherapy may be delayed by 1-3 days if clinically indicated.
  Other Names: Fludara®; Fludarabine phosphate; 2-fluoro-ara-AMP
Drug: Cytarabine — Will be given IV over 4 hours daily on days 16 through 20. Cytarabine may be given prior to day 16 if it is determined to be in the participant's best interest based on disease progression. Chemotherapy may be delayed by 1-3 days if clinically indicated.
  Other Names: Cytosine arabinoside; Ara-C; Cytosar®
Drug: methotrexate/hydrocortisone/cytarabine — Intrathecal (IT) triples will be given prior to cycle 1: IT cytarabine, IT methotrexate, and IT methotrexate/hydrocortisone/cytarabine (MHA) are acceptable. Patients without evidence of central nervous system (CNS) leukemia will receive no further IT therapy during cycle 1. Patients with CNS disease will receive weekly ITMHA until the cerebrospinal fluid becomes free of leukemia (minimum of 4 doses).
  Other Names: ITMHA; Intrathecal triples

SUMMARY:
The purpose of this study is to test the safety of selinexor (KPT-330) and to find the highest dose of selinexor (KPT-330) that can be given safely when it is combined with two chemotherapy drugs (fludarabine and cytarabine). This study will be done in two parts: Phase I and Phase II.

The goal of Phase I is to find the highest tolerable dose of selinexor (KPT-330) that we can give to patients with leukemia or MDS, when it is combined with fludarabine and cytarabine.

The goal of the subsequent Phase II portion of the study (insert NCT ID of SELHEM-2) is to give the highest dose of selinexor (KPT-330) in combination with fludarabine/cytarabine that was found in Phase I to be safe for children with leukemia or MDS. The investigators will examine the effect of this combination treatment.

PRIMARY OBJECTIVE:

* Determine a tolerable combination of selinexor, fludarabine, and cytarabine in pediatric patients with relapsed or refractory hematologic malignancies included acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), mixed phenotype acute leukemia (MPAL) and myelodysplastic syndrome (MDS).

SECONDARY OBJECTIVES:

* To characterize the pharmacokinetics of selinexor, when administered in tablet form, after the first dose and at steady-state, as well as in combination with fludarabine and cytarabine
* To estimate the overall response rate of selinexor given with fludarabine and cytarabine in patients with relapsed or refractory hematologic malignancies

DETAILED DESCRIPTION:
Phase I will characterize the dose-limiting toxicities (DLTs) and determine the maximum tolerated dose (MTD) or recommended phase II dose of selinexor when given in combination with fludarabine and cytarabine.

Selinexor will be given twice weekly (on days 1 and 3) and escalated or de-escalated based on tolerability. The rolling-6 design will be used for this study. Only cycle 1 of therapy will be used to evaluate the DLT. Two to six participants can be concurrently enrolled onto a dose level, dependent on 1) the number of participants enrolled at the current dose level, 2) the number of participants who have experienced DLT at the current dose level, and 3) the number of participants entered but with tolerability data pending at the current dose level. Accrual is suspended when a cohort of six has enrolled or when the study endpoints have been met.

Once the recommended Phase II dose is determined, additional patients will be enrolled, if necessary, so that at least 6 subjects are treated with the recommended Phase II dose to determine MTD. After the MTD is determined, 12 additional patients will be treated at this dose level for further evaluation of tolerability and response.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of AML, MDS, ALL or MPAL and must have disease that has relapsed or is refractory to chemotherapy, or that has relapsed after hematopoietic stem cell transplantation (HSCT)

  * Refractory disease is defined as persistent disease after at least two courses of induction chemotherapy.
  * Patients with AML, MPAL or MDS are eligible at first or subsequent relapse, whereas patients with ALL are eligible at second or subsequent relapse or any relapse that is refractory to salvage chemotherapy.
  * Patients with AML or ALL must have ≥ 5% leukemic blasts in the bone marrow or increasing levels of MRD in the bone marrow as assessed by flow cytometry. If an adequate bone marrow sample cannot be obtained, patients may be enrolled if there is unequivocal evidence of leukemia in the peripheral blood.
* Adequate organ function defined as the following:

  * Direct bilirubin ≤ 1.5 x institutional upper limit of normal (IULN)
  * AST (SGOT)/ALT (SGPT) < 3 x IULN
  * Creatinine within normal institutional limits for age
* Prothrombin time (PT) and partial thromboplastin (PTT) ≤ 1.5 x IULN.
* Age criteria: Patients treated at collaborating sites and current St. Jude patients who are on therapy or within 3 years of completion of therapy must be ≤ 24 years old. All other St. Jude patients must be < 21 years old.
* Patients must be able to swallow tablets.
* Performance status: Lansky ≥ 50 for patients who are ≤ 16 years old and Karnofsky ≥ 50% for patients who are > 16 years old.
* Patients must have fully recovered from the acute effects of all prior therapy.
* For patients who have received prior HSCT, there can be no evidence of GVHD and greater than 60 days must have elapsed since the HSCT.

Exclusion Criteria:

* History of cerebellar toxicity or cerebellar neurological findings on exam.
* Must not be pregnant or breastfeeding. Female patients of child-bearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test at screening, and male patients must use an effective barrier method of contraception if sexually active with a female of child-bearing potential. Acceptable methods of contraception are condoms with contraceptive foam, oral, implantable or injectable contraceptives, contraceptive patch, intrauterine device, diaphragm with spermicidal gel, or a sexual partner who is surgically sterilized or post-menopausal. For both male and female patients, effective methods of contraception must be used throughout the study and for three months following the last dose.
* Patients with Down syndrome, acute promyelocytic leukemia, juvenile myelomonocytic leukemia, Fanconi anemia, Kostmann syndrome, Shwachman syndrome, or other bone marrow failure syndromes are not eligible.
* Use of investigational agents, with the exception of gemtuzumab ozogamicin, within 30 days.
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, study participation, follow up, or interpretation of study research.
* Unstable cardiovascular function:

  * symptomatic ischemia
  * congestive heart failure NYHA Class > 3
  * myocardial infarction (MI) within 3 months
* Uncontrolled infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to first dose. Infections controlled on concurrent anti-microbial agents are acceptable, and anti-microbial prophylaxis per institutional guidelines are acceptable.
* Known human immunodeficiency virus (HIV) infection (pre-study testing not required).
* Patients with malabsorption syndrome, or any other disease significantly affecting gastrointestinal function.
* Prior treatment with selinexor.

Max Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of combination selinexor, fludarabine and cytarabine | MTD will be determined at the end of cycle 1 (day 35 of therapy)
  The MTD is empirically defined as the highest dose level at which six participants have been treated with at most one participant experiencing a DLT and the next higher dose has been determined to be too toxic. If the lowest dose level studied is too toxic or the highest dose level studied is considered safe, the MTD will not have been considered estimated.
Dose limiting toxicity of combination selinexor, fludarabine and cytarabine | During cycle 1 of therapy (days 1-35)
  Any participant who experiences dose-limiting toxicities (DLT) at any time during the first 35 days after taking the initial dose of selinexor and before receiving non-protocol therapy (such as transplant) is considered evaluable for toxicity. Participants without DLT who receive at least 5 of the 6 prescribed cycle I doses of selinexor and can be followed for 35 days following their initial dose of selinexor are also considered evaluable for toxicity. Participants who are not evaluable for toxicity (such as those removed early from therapy to start alternate therapy) at a given dose level will be replaced.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of selinexor | Days 1-3 (pre-dose, 30 minutes, and 1, 2, 4, 8, 24, and 48 hours after dose) and Day 22 (pre-dose and 1, 2, 4, and 8 hours after day 22 dose)
  The pharmacokinetics of selinexor as well as selinexor in combination with fludarabine and cytarabine will be determined.
  Plasma samples will be analyzed for selinexor concentration. Selinexor concentration data will be analyzed in a non-linear mixed effects population PK model with potential covariates including age, body weight, gender, disease state, hepatic or renal function, concomitant medications, and treatment. Details of the population PK analysis, including software, post-processing and statistical analysis, will be outlined in a separate Data Analysis Plan. Interim analysis may be conducted on plasma selinexor concentration data throughout the study. Summary statistics, including mean, median, standard deviation, coefficient of variation and group size may be compiled and reported during the study. Interim analysis of PK parameters and biomarker analyses may be performed in order to provide a pharmacokinetic-pharmacodynamic assessment throughout the study.
complete response rate | between days 28 and 35 of cycle 1
  The efficacy of the combination of selinexor, fludarabine, and cytarabine, as measured by the complete response (CR) rate and the overall response (OR) rate (CR + CRi + PR) will be assessed for the patients enrolled at the MTD. The rates of CR and OR will be presented as a point estimate with a 95% exact binomial confidence interval.
Overall response rate | Between days 28 and 35 of cycle 1
  The efficacy of the combination of selinexor, fludarabine, and cytarabine, as measured by the complete response (CR) rate and the overall response (OR) rate (CR + CRi + PR) will be assessed for the patients enrolled at the MTD. The rates of CR and OR will be presented as a point estimate with a 95% exact binomial confidence interval.
Area under the curve (AUC) of selinexor | Days 1-3 (pre-dose, 30 minutes, and 1, 2, 4, 8, 24, and 48 hours after dose) and Day 22 (pre-dose and 1, 2, 4, and 8 hours after day 22 dose)
  The pharmacokinetics of selinexor as well as selinexor in combination with fludarabine and cytarabine will be determined.
  Plasma samples will be analyzed for selinexor concentration. Selinexor concentration data will be analyzed in a non-linear mixed effects population PK model with potential covariates including age, body weight, gender, disease state, hepatic or renal function, concomitant medications, and treatment. Details of the population PK analysis, including software, post-processing and statistical analysis, will be outlined in a separate Data Analysis Plan. Interim analysis may be conducted on plasma selinexor concentration data throughout the study. Summary statistics, including mean, median, standard deviation, coefficient of variation and group size may be compiled and reported during the study. Interim analysis of PK parameters and biomarker analyses may be performed in order to provide a pharmacokinetic-pharmacodynamic assessment throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey E. Rubnitz, MD,PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (6):
- United States (6):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of Chicago, Chicago, Illinois
  - Duke University Medical Center, Durham, North Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas

REFERENCES:
- [Result] Alexander TB, Lacayo NJ, Choi JK, Ribeiro RC, Pui CH, Rubnitz JE. Phase I Study of Selinexor, a Selective Inhibitor of Nuclear Export, in Combination With Fludarabine and Cytarabine, in Pediatric Relapsed or Refractory Acute Leukemia. J Clin Oncol. 2016 Dec;34(34):4094-4101. doi: 10.1200/JCO.2016.67.5066. Epub 2016 Oct 31. PMID 27507877
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols